CLINICAL TRIAL: NCT07140874
Title: Evaluation of Supplemental Zinc as an Adjunct to Prolong the Duration of Benefit After Botulinum Toxin Injections in Subjects With Cervical Dystonia
Brief Title: Zinc as an Adjunctive Therapy for Cervical Dystonia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB202500431
Record Dates: First submitted 2025-08-15; First posted 2025-08-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-08

CONDITIONS: Cervical Dystonia
Keywords: cervical dystonia; botulinum toxin; Botox; zinc citrate; zinc
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zinc first (Experimental): Encapsulated zinc citrate 30 mg orally daily for 3 months followed by placebo capsule matching zinc daily for 3 months
  Interventions: Drug: Zinc citrate; Drug: Placebo
- Placebo first (Experimental): Placebo capsule matching zinc daily for 3 months, followed by encapsulated zinc citrate 30 mg orally daily for 3 months
  Interventions: Drug: Zinc citrate; Drug: Placebo

INTERVENTIONS:
Drug: Zinc citrate — Oral zinc citrate 30 mg daily
Drug: Placebo — Placebo

SUMMARY:
The goal of this clinical trial is to evaluate if supplemental zinc can prolong the duration of benefit of botulinum toxin injections in cervical dystonia patients receiving care at the University of Florida.

The main aims are:

1. To evaluate the efficacy of zinc citrate supplementation in prolonging the duration of symptom relief provided by botulinum toxin type A (Botox) injections in cervical dystonia patients.
2. To assess the safety and tolerability of zinc supplementation in this patient population.
3. To analyze the potential influence of zinc supplementation on the quality of life and functional outcomes in cervical dystonia patients receiving Botox.

Researchers will compare zinc citrate to a placebo (a look-alike substance that contains no active drug) to see if zinc works to extend the effects of Botox.

Participants will:

Take zinc citrate or a placebo every day for 3 months, then cross over to the alternative treatment for another 3 months.

Visit the clinic every 3 months for Botox injections, check ups and surveys.

DETAILED DESCRIPTION:
Study Design:

* Randomized, single-blind, crossover placebo-controlled trial.
* Participants: Approximately 20 patients diagnosed with cervical dystonia and currently receiving botulinum toxin (BoNT) type A (Botox) injections at the University of Florida (UF) Movement Disorders Clinic with good response to treatment as determined by treating neurologist will be enrolled into this study. The investigators plan to screen 25 patients to allow for screen failures and withdrawals.
* Intervention: Participants will be randomized to receive either zinc citrate 30 mg supplementation or placebo starting immediately after their scheduled BoNT injection for 3 months. At a follow up BoNT injection, they will receive the alternative treatment for another 3 months. The total observation period is 6 months. Standard time between BoNT injections is 3 months.

The UF Movement Disorders Clinic follows approximately 1,500 cervical dystonia patients a year. The investigators do not anticipate any recruitment challenges.

Participants will be recruited during neurology clinic appointments and screening clinic appointments.

* Patients will receive the same pattern of BoNT injections (muscle selection and dose) during the duration of the study.
* Blood serum levels of zinc and vitamin B12 and complete blood counts (CBCs) will be measured at baseline and at the end of the study. Participants will be sent to UF Health Medical lab for blood draws and sample collection.
* Written informed consent will be obtained from each participant before any study-specific procedures or assessments are performed.

Inclusion Criteria:

* Adults aged 18-65 years.
* Diagnosed with cervical dystonia.
* Receiving regular BoNT type A (Botox) injections for at least one year.

Exclusion Criteria:

* Known allergy or intolerance to zinc.
* Significant comorbidities or concurrent medications that could interfere with study outcomes.
* Pregnant or breastfeeding women.
* Already taking a zinc supplement which would exceed tolerable upper intake level in adults (40 mg elemental zinc per day) with addition of zinc study supplement

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years.
* Diagnosed with cervical dystonia.
* Receiving regular BoNT type A (Botox) injections for at least one year.

Exclusion Criteria:

* Known allergy or intolerance to zinc.
* Significant comorbidities or concurrent medications that could interfere with study outcomes.
* Pregnant or breastfeeding women.
* Already taking a zinc supplement which would exceed tolerable upper intake level in adults (40 mg elemental zinc per day) with addition of zinc study supplement.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration of Botox efficacy | 3 and 6 month post intervention
  Time to return to baseline symptom severity using the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Severity Subscale. The TWSTRS Severity Subscale is scored from 0 to 35, with higher numbers indicating a more severe condition.

SECONDARY OUTCOMES:
Change in Pain Severity at 3 months | 3 months post intervention
  Change in pain severity at 3 months as measured by the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Pain Subscale. The TWSTRS Pain Subscale is scored from 0 to 20, with higher numbers indicating a more painful condition.
Change in Quality of Life at 3 months | 3 months post intervention
  Change in quality of life at 3 months as measured by the Craniocervical dystonia questionnaire (CDQ-24). The CDQ-24 contains 24 items pertaining to quality of life in patients with cervical dystonia, scored from 0 ("never") to 4 ("very severely").
Change in Functional Disability at 3 months | 3 months post intervention
  Change in functional disability at 3 months as measured by the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) Disability Subscale. The TWSTRS Disability Subscale is scored from 0 to 30 with higher numbers indicating a more disabling condition.
Patient Global Impression of Change | 3 months post intervention
  Patient Global Impression of Change (PGIC) at 3 months. The PGIC measures the patient's perception of the change in their condition after treatment, scored from 1 ("Very much improved") to 7 ("Very much worse").
Clinician Global Impression of Change | 3 months post intervention
  Clinician Global Impression of Change (CGIC) at 3 months. The CGIC measures the researcher's perception of the change in the patient's condition after treatment, scored from 1 ("Very much improved") to 7 ("Very much worse").

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Fanty, MD, Principal Investigator — University of Florida
Locations (1):
- Norman Fixel Institute for Neurological Diseases, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Study researchers will be performing the analysis

REFERENCES:
- [Background] Betul Ergul A, Turanoglu C, Karakukcu C, Guler Kazanci E, Altuner Torun Y. Increased vitamin B12 levels in children with zinc deficiency. Int J Vitam Nutr Res. 2017 Sep;87(5-6):247-252. doi: 10.1024/0300-9831/a000444. Epub 2018 Aug 10. PMID 30095365
- [Background] Rabinovich D, Smadi Y. Zinc. 2023 May 1. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK547698/ PMID 31613478
- [Background] Shemais N, Elarab AE, ElNahass H. The effect of botulinum toxin A in patients with excessive gingival display with and without zinc supplementation: randomized clinical trial. Clin Oral Investig. 2021 Nov;25(11):6403-6417. doi: 10.1007/s00784-021-03944-2. Epub 2021 May 5. PMID 33950373
- [Background] Jeng SS, Chen YH. Association of Zinc with Anemia. Nutrients. 2022 Nov 20;14(22):4918. doi: 10.3390/nu14224918. PMID 36432604
- [Background] Junior HT, dos Santos Melo C, Mendes RR et al. Effects of zinc supplementation on duration and action of botulinum toxin applied to face muscles: A systematic review of randomized clinical trials. Journal of Trace Elements and Minerals. 5. 100080. 10.1016/j.jtemin.2023.100080.
- [Background] Xing Y, O'Suilleabhain P. Does Oral Zinc Supplementation Augment the Effect of Botulinum Neurotoxin in Dystonia? Neurology 2015;84(14 Supplement):P4.330. doi: 10.1212/WNL.84.14_supplement.P4.330
- [Background] Mallat F, Kaikati J, Kechichian E. Botulinum Toxins and Zinc: From Theory to Practice-A Systematic Review. Clin Neuropharmacol. 2023 Jun 20. doi: 10.1097/WNF.0000000000000557. Online ahead of print. PMID 37335837
- [Background] Koshy JC, Sharabi SE, Feldman EM, Hollier LH Jr, Patrinely JR, Soparkar CN. Effect of dietary zinc and phytase supplementation on botulinum toxin treatments. J Drugs Dermatol. 2012 Apr;11(4):507-12. PMID 22453589